CLINICAL TRIAL: NCT06837740
Title: The Effects of Music Therapy and Aromatherapy Interventions on Pulse Rate, Blood Pressure, Anxiety, and Self-Esteem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, Hediye Utli, PhD, RN, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: hediyee
Record Dates: First submitted 2025-02-05; First posted 2025-02-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Aromatherapy; Music Therapy
Keywords: Pulse Rate; Blood Pressure; Anxiety; Self-Esteem
MeSH Terms: conditions — Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: Aromatherapy group Aromatherapy with music therapy group Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy group (Experimental): Experimental
  Interventions: Other: Aromatherapy group
- Aromatherapy with music therapy group (Active Comparator): Active comparator
  Interventions: Other: Aromatherapy with music therapy group
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: Aromatherapy group — Effects of Aromatherapy Interventions
  Arms: Aromatherapy group
Other: Aromatherapy with music therapy group — Effects of Music Therapy and Aromatherapy Interventions
  Arms: Aromatherapy with music therapy group

SUMMARY:
Appropriate intervention methods should be investigated to reduce stress and fatigue of students in psychomotor skills. The aim of this study is to reveal the effects of music therapy and aromatherapy interventions on pulse, blood pressure, anxiety and self-esteem levels of nursing students during injection application to the ventrogluteal region on a mannequin.

Hypotheses:

H1a= During the ventrogluteal injection application of nursing students on a mannequin, Aromatherapy and Music therapy and Aromatherapy application have an effect on pulse rate.

H1b= During the ventrogluteal injection application of nursing students on a mannequin, Aromatherapy and Music therapy and Aromatherapy application have an effect on blood pressure level.

H1c= During the ventrogluteal injection application of nursing students on a mannequin, Aromatherapy and Music therapy and Aromatherapy application have an effect on anxiety level.

H1d= During the ventrogluteal injection application of nursing students on a mannequin, Aromatherapy and Music therapy and Aromatherapy application have an effect on self-esteem level.

DETAILED DESCRIPTION:
Appropriate intervention methods should be investigated to reduce stress and relieve fatigue of students in psychomotor skills. The aim of this study is to reveal the effects of Music therapy and Aromatherapy interventions on pulse, blood pressure, fatigue and self-esteem levels of nursing students during ventrogluteal injection application. For this purpose, the investigators tried to provide more information to the literature for Music therapy and Aromatherapy interventions in this single-blind randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Students who are first year students, and
* Volunteer to participate in the research will be included.

Exclusion Criteria:

* Volunteer to participate in the research will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Pulse Rate | "Average of 1 year"
  Pulse Rate
Systolic and Diastolic Pressure | "Average of 1 year"
  Systolic and Diastolic Pressure
Anxiety | "Average of 1 year"
  State Anxiety Inventory: It has also been translated and adapted into Turkish by Oner and Le Compte. It is a measurement tool consisting of statements indicating how a person feels at a certain moment.
Self-Esteem | "Average of 1 year"
  Rosenberg Self-Esteem Scale Form: The scale, developed by Rosenberg to measure self-esteem, was adapted into Turkish by Çuhadaroğlu.

CONTACTS AND LOCATIONS:
Overall Officials: Hediye Utli, PhD, Study Director — Mardin Artuklu University
Locations (1):
- a university in eastern Turkey, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No